CLINICAL TRIAL: NCT02691117
Title: Topical Garlic Concentrate for Alopecia Areata in Children: A Prospective Open Label Study
Brief Title: Topical Garlic Concentrate for Alopecia Areata in Children
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy of the study medication
Sponsor: Elena Pope (Other)
Collaborators: Dermatology Foundation (Other)
Responsible Party: Sponsor-Investigator, Elena Pope, Professor of Paediatrics, University of Toronto Fellowship Director and Section Head, Paediatric Dermatology, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000050555
Record Dates: First submitted 2015-12-15; First posted 2016-02-25 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata; Garlic concentrate
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Garlic concentrate (Experimental): Garlic gel concentrate- once a day topical application
  Interventions: Drug: garlic concentrate

INTERVENTIONS:
Drug: garlic concentrate — Topical application of GarlicRich gel on the scalp areas affected with alopecia areata once a day for 6 months
  Other Names: GarlicRich

SUMMARY:
Management of pediatric alopecia is particularly challenging given the chronicity of the condition, limited therapeutic response and devastating psychological effects. There is a paucity of safe and effective therapies in this population.

The investigators propose to conduct and open label, prospective cohort pilot study using topical garlic concentrate ( GarlicRich) for treatment of children with alopecia areata. Study medication will be applied topically on affected area of the skin daily for 6 months. Follow up visits will occur monthly to access the efficacy and safety of the proposed treatment .

DETAILED DESCRIPTION:
The investigators are planning to enroll in the study 20 participants at Sickkids.

It is an open label, prospective cohort pilot study. Patients enrolled in the study will be followed at the Hospital for Sick Children for 6 months. Participants will come for the study visits every month (7 study visits). During each study visit two investigators will independently access patient's hair density and calculate the SALT score (Severity of Alopecia Tool Score), using the participant's digital photographs.

Patients will be provided with the study medication for all duration of the study.

The results of the treatment will be compared with the baseline data ( pictures/ scores/ hair density) to evaluate the efficacy and safety of garlic concentrate in children with patchy alopecia areata.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 years and older up to 18 years of age
* Patches of alopecia areata that affect less than 50% of the scalp.
* Alopecia of at least 1 year duration without evidence of regrowth
* Informed written consent

Exclusion Criteria:

* Any children experiencing significant spontaneous regrowth of terminal hair at the baseline visit.
* Any children treated with a topical, (including shampoos with active ingredients like minoxidil or clobetasol), intralesional or systemic agent likely to cause regrowth in alopecia areata within the past month from the baseline visit and during study period.
* Children with history of hypersensitivity to garlic.
* Children with widespread alopecia areata as alopecia totalis, universalis, ophiasis or diffuse Alopecia Areata.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Percentage change of SALT scores at 6 months compared to baseline. | 6 months
  Percentage change of SALT scores at 6 months compared to baseline

SECONDARY OUTCOMES:
Categorical percent hair regrowth | 6 months
  SALT derived percent regrowth, categorized as: A0 = no change or further loss; A1= 1-24% regrowth; A2= 25-49% regrowth; A3= 50-74% regrowth; A4= 75-99% regrowth; A5= 100% regrowth
Proportion of subjects with at least 70% hair regrowth using the percent scalp hair regrowth based on SALT score. | 6 months
  Proportion of subjects with at least 70% hair regrowth using the percent scalp hair regrowth based on SALT score.
Density of hair regrowth at 6 months | 6 months
  Density will be measured by using a dermatoscope and calculating the number of hairs in the field
Type of hair regrowth at 6 months | 6 months
  Type of hair will be a categorical variable with 3 types of values: vellus, indeterminate and terminal hairs
Parental/patient assessment of hair regrowth using a 100 mm visual analog scale with 3 anchors (total loss, no change, full regrowth) where 5 mm corresponds to 10% change | 6 months
  VOS will be used by parents/ patient only once at the final study visit to access the result of the study treatment.
Intra-class correlations between the two investigators' assessments using SALT and VAS assessment of hair regrowth | 1,2,3,4,5,6 months
  The results of two study investigator's assessment (SALT and VAS) will be compared at each study visit.
Correlation between surface area and SALT score | 1,2,3,4,5,6 months
  Correlation between surface area and SALT score
Correlation between SALT scores and parental/patient assessment of regrowth at 6 months. | 6 months
  Correlation between SALT scores and parental/patient assessment of regrowth
Percentage of patients experiencing adverse effects (erythema, irritation, contact dermatitis), collected by investigator and reported by the parents in the study diaries. | 0-6 months
  Percentage of patients experiencing adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Elena Pope, MD, MSc, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Th Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
only aggregated data will be available to participants